CLINICAL TRIAL: NCT01002079
Title: A Study of the Effect of Concomitant Administration of Rifampin on the Pharmacokinetics of BMS-708163 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study With Rifampin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CN156-028
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BMS-708163 (Experimental)
  Interventions: Drug: BMS-708163
- Rifampin (Other)
  Interventions: Drug: Rifampin
- Rifampin + BMS-708163 (Experimental)
  Interventions: Drug: BMS-708163; Drug: Rifampin

INTERVENTIONS:
Drug: BMS-708163 — Capsule, Oral, 125 mg, Once daily, 1 day
  Arms: BMS-708163; Rifampin + BMS-708163
Drug: Rifampin — Capsule, Oral, 600 mg, Once daily, 7 days
  Arms: Rifampin
Drug: Rifampin — Capsule, Oral, 600 mg, Once daily, 6 days
  Arms: Rifampin + BMS-708163

SUMMARY:
The purpose of the study is to determine if the concomitant administration of rifampin with BMS-708163 will affect the Pharmacokinetics of BMS-708163 and to assess safety and tolerability of co-administration BMS-708163 and rifampin

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and postmenopausal female subjects, 18-55 yrs old inclusive

Exclusion Criteria:

* Women of childbearing potential
* Tuberculosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
BMS-708163 alone and with rifampin: BMS-708163 single dose PK parameters (Cmax, Tmax, T-HALF, AUC(0-T), AUC(INF), CLT/F and molar AUCmet/AUCparent ratios will be assessed without rifampin (Day 1) and with rifampin (Day 13) | Within 30 days after dose

SECONDARY OUTCOMES:
BMS-708163 alone and with rifampin: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Within 30 days after dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Bangalore, India

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx